CLINICAL TRIAL: NCT05392140
Title: The Effect of Smart Phone Application Supported Nursing Care Program on the Self-Management of Hypertensive Patients
Brief Title: The Effect of Smart Phone Application Supported Nursing Care Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kastamonu University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Zeynep Arabacı, lecturer, Kastamonu University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: no sponsors
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hypertension
Keywords: Nursing, Medication adherence, Hypertension
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The research was organized in an experimental design with pre-test post-test control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group. (Experimental): Health belief model-based smartphone-assisted nursing care program application will be installed on the phones of the patients who will be in the intervention group.
  Interventions: Behavioral: Health belief model-based smartphone-assisted nursing care program application will be installed on the phones of the patients who will be in the intervention group.
- non-intervention group (Active Comparator): standard care practice will continue
  Interventions: Behavioral: Standart care

INTERVENTIONS:
Behavioral: Health belief model-based smartphone-assisted nursing care program application will be installed on the phones of the patients who will be in the intervention group. — Health belief model-based smartphone-assisted nursing care program application will be installed on the phones of the patients who will be in the intervention group.
  Arms: intervention group.
Behavioral: Standart care — Standart care
  Arms: non-intervention group

SUMMARY:
Hypertension is an important public health problem in our country and in the world. For success in hypertension treatment, timely and accurate diagnosis of patients, effective implementation of lifestyle changes, timely initiation of drug therapy and effective drug compliance are emphasized. The rapid adoption of smartphone technology provides a promising platform for overcoming drug non-compliance by providing medication intake reminders, healthy lifestyle education. It is emphasized that the health belief model can be used in the self-management of the hypertension patient's health and in the regulation of services with smart phone applications. Based on these facts, this study was planned to examine the effect of the smart phone management system supported nursing care program given by the nurse to the primary hypertension patients registered in the Family Health Center on the patient's compliance with the treatment and the blood pressure staying within the target limits. The research was organized in an experimental design with pre-test post-test control group. The population of the research consists of primary hypertensive patients registered in Family Health Centers in Tosya district of Kastamonu province. It is planned to include a total of 102 people, 51 in the intervention and control groups, in the sample group.

DETAILED DESCRIPTION:
Hypertension is an important public health problem in our country and in the world. For success in hypertension treatment, timely and accurate diagnosis of patients, effective implementation of lifestyle changes, timely initiation of drug therapy and effective drug compliance are emphasized. The rapid adoption of smartphone technology provides a promising platform for overcoming drug non-compliance by providing medication intake reminders, healthy lifestyle education. It is emphasized that the health belief model can be used in the self-management of the hypertension patient's health and in the regulation of services with smart phone applications. Based on these facts, this study was planned to examine the effect of the smart phone management system supported nursing care program given by the nurse to the primary hypertension patients registered in the Family Health Center on the patient's compliance with the treatment and the blood pressure staying within the target limits. The research was organized in an experimental design with pre-test post-test control group. The population of the research consists of primary hypertensive patients registered in Family Health Centers in Tosya district of Kastamonu province. Sample, effect size 0.25; By taking the alpha value of 0.05 and the power of 0.80, the minimum number of samples was calculated as 82. Considering that there may be data losses, it is planned to include a total of 102 people, 51 in the intervention and control groups, in the sample group. In data collection, the "Patient Information Form", "Blood pressure follow-up form" prepared by the researcher, and the adaptation to Turkish will be collected with the help of the "Drug Adherence/Compliance Self-Efficacy Scale" prepared by Gözüm and Hacıhasanoğlu in 2005. Health belief model-based smartphone-assisted nursing care program application will be installed on the phones of the patients who will be in the intervention group. After the application is started to be used, patients will be notified every two weeks for six months for the disease management process to have nutrition, exercise and doctor control processes. Patients will be able to send a message to the nurse through the application. Messages will be answered regularly on a designated day each week. The data will be collected by face-to-face interview method after necessary explanations and necessary consents are obtained by the researchers. One month after the posttest application (second data), application predicate and usage, the third data (1st follow-up) will be collected in the 3rd month, the fourth data (2nd follow-up) will be collected in the 6th month.

ELIGIBILITY:
Inclusion Criteria:

* -Agreeing to participate in the research.
* Being between 45-64 years old
* At least primary school graduate
* Using antihypertensive medication for at least 6 months with the diagnosis of primary (essential) hypertension.
* Owning a smart phone

Exclusion Criteria:

* Being diagnosed with secondary hypertension Have been diagnosed with pregnancy-onset hypertension
* Hearing, seeing and understanding problems Having a diagnosis of dementia and alzheimer's
* Diagnosed with chronic kidney failure
* Being a dialysis patient
* History of myocardial infarction, stroke, diagnosis of heart failure

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
There is a difference in time (pre-test, after intervention, 1st month, 3rd month, 6th month) between intervention and control group patients' self-efficacy scale scores of adherence to drug therapy. | 0-6 month
  Drug Adherence/Compliance Self-Efficacy Scale

SECONDARY OUTCOMES:
There is a difference in time (pre-test, after the intervention, 1st month, 3rd month, 6th month) between the patients in the intervention and control groups having normal systolic and diastolic blood pressure measurements. | 0-6 month
  Blood pressure follow-up form

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ARABACI, Study Chair — Kastamonu University

IPD SHARING:
Plan to Share IPD: No